CLINICAL TRIAL: NCT04339868
Title: Terlipressin Versus Placebo for Septic Shock Refractory to High Doses Catecholamine Vasopressors: A Randomized-controlled Trial
Brief Title: Terlipressin for Refractory Septic Shock
Acronym: TERESEP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si 049/2020
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Septic Shock; Refractory Shock; Norepinephrine Adverse Reaction
MeSH Terms: conditions — Shock, Septic; Shock | interventions — Terlipressin

STUDY DESIGN:
Intervention Model Description: Intervention arm: Terlipressin plus Norepinephrine and/or Epinephrine Controlled arm: Placebo plus Norepinephrine and/or Epinephrine for Treatment Refractory Septic Shock
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Performed a randomization table before enrollment. Prepare the study drug receiving or placebo receiving according to sequential number derived from the randomization table and keep it in a conceal envelop. Prepare study drug and placebo by a pharmacist or an investigation nurse, according to the randomization table number, and keep both study drug and placebo in the identical containment which labeled by a sequential number. Once a patient was enrolled and informed was signed, then study drug or placebo was start according to sequential number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terlipressin group (Active Comparator): Terlipressin acetate 1 mg in 0.9% normal saline (NaCl) 50 mL (0.02 mg/mL) Initial dose 20 mcg/hr (1 mL/hr) titrate increase 1 mL/hr every 30 min to 100 mcg/hr (5 mg/hr) to keep mean arterial blood pressure (MAP) > 65 mmHg If MAP > 75 mmHg for > 30 min, decrease epinephrine and norepinephrine until < 0.15 mcg/kg/min, then decrease terlipressin until stop
  Interventions: Drug: Terlipressin
- Placebo group (Placebo Comparator): Placebo 0.9% NaCl 50 mL Initial dose 1 mL/hr titrate increase 1 mL/hr every 30 min to 5 mg/hr to keep mean arterial blood pressure (MAP) > 65 mmHg If MAP > 75 mmHg for > 30 min, decrease epinephrine and norepinephrine until < 0.15 mcg/kg/min, then decrease placebo until stop
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Terlipressin — Terlipressin (20-100 mcg/hr) plus norepinephrine and/or epinephrine
  Arms: Terlipressin group
Drug: Placebo — 0.9% NaCl plus norepinephrine and/or epinephrine
  Arms: Placebo group

SUMMARY:
Norepinephrine was recommended as the first vasopressor for septic shock resuscitation.

For the patient who did not response to high dose norepinephrine, epinephrine was recommended.

Vasopressin was also recommended as an alternative vasopressor, in case patient did not response to norepinephrine and or epinephrine.

Terlipressin, a selective V1 receptor binding with long half life, was reported that it main action is to increase blood pressure via the different mechanism from norepinephrine and epinephrine.

To use terlipressin, combine with norepinephrine and or epinephrine among refractory septic shock, could decrease the usage dose of norepinephrine and epinephrine as well as lower the side effects of too high adrenergic stimuli.

DETAILED DESCRIPTION:
Norepinephrine was recommended as the first vasopressor for septic shock resuscitation.

For the patient who did not response to high dose norepinephrine, epinephrine was recommended.

Both norepinephrine and epinephrine action via the alpha adrenergic stimuli to increase vascular smooth muscle contraction, induced vasoconstriction and increase arterial blood pressure. It also action via beta adrenergic stimuli, to increase heart rate and myocardial contractility, then increase stroke volume and cardiac output.

Too much alpha and beta adrenergic stimulation, especially during received high dose norepinephrine and or epinephrine associated with vasoconstriction induce organs ischemia.

The most common organ ischemia included myocardial ischemia, bowel ischemia and limbs ischemia.

Cardiac arrhythmia was also the most common complication associated with high dose norepinephrine and or epinephrine.

Atrial fibrillation was the most common reported arrhythmia, however, fatal arrhythmia included ventricular fibrillation and tachycardia were also reported.

Vasopressin was recommended as an alternative vasopressor, in case patient did not response to norepinephrine and or epinephrine.

Terlipressin, a selective V1 receptor binding with long half life, was reported that it main action is to increase blood pressure via the different mechanism from norepinephrine and epinephrine.

To use terlipressin, combine with norepinephrine and or epinephrine among refractory septic shock, could decrease the usage dose of norepinephrine and epinephrine as well as lower the side effects of too high adrenergic stimuli.

The benefit effect of terlipressin could be demonstrated when prescribe among the septic shock patients who required high dose of adrenergic vasoactive agents.

Terlipressin plus norepinephrine and or epinephrine could maintain or even improve blood pressure and tissue perfusion with lower fatal side effects than norepinephrine and or epinephrine without terlipressin.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock according to Sepsis-3 definition
* Evidence of adequate fluid
* Received norepinephrine 0.2 mcg/kg/min or more
* Received norepinephrine plus epinephrine (any dose)
* Mean arterial lower than 65 mmHg or lactate > 2 mmol/liter

Exclusion Criteria:

1. Septic shock diagnosis > 48 hours before
2. Receive intravenous fluid < 30 mL/kg before enrollment
3. Do-not-resuscitation and terminally ill
4. Refractory to treatment malignancy
5. Pregnancy

7. Chronic renal failure stage 5 with no plan for long term renal replacement therapy 8. Cirrhosis child C 9. Cardiogenic shock 10. Acute decompensated heart failure 11. Evidence of left ventricular ejection fraction (LVEF) < 35% 12. Acute coronary syndrome within 72 hours 13. Severe valvular heart disease 14. Documented life-threatening tachyarrhythmia before enrollment 15. Diagnosis of acute mesenteric ischemia before enrollment 16. Previous diagnosis of Raynaud's phenomenon 17. Known peripheral arterial disease 18. Refuse to sign the informed consent by patient or representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Achieve target blood pressure with low dose adrenergic agents | 6 hours after initiate study drug
  Achieve target mean arterial blood pressure 65 millimeter mercury or more with norepinephrine and/or epinephrine dose 0.2 mcg/kg/min or lower

SECONDARY OUTCOMES:
28 day mortality | 28 days
  Proportion of patient who dead before 28 days after enrollment
Mean arterial blood pressure | 72 hours
  Mean arterial blood pressure after initiate study drug
Hospital mortality | 90 days
  Proportion of patient who dead before hospital discharge after enrollment
ICU mortality | 90 days
  Proportion of patient who dead before ICU discharge after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Surat Tongyoo, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Medicine, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
The data set and analysis are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After complete enrollment and for 24 months
Access Criteria: Please direct contact to the principle investigator

REFERENCES:
- [Result] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Permpikul C, Tongyoo S, Viarasilpa T, Trainarongsakul T, Chakorn T, Udompanturak S. Early Use of Norepinephrine in Septic Shock Resuscitation (CENSER). A Randomized Trial. Am J Respir Crit Care Med. 2019 May 1;199(9):1097-1105. doi: 10.1164/rccm.201806-1034OC. PMID 30704260